CLINICAL TRIAL: NCT06309862
Title: Association of Immune Checkpoint Inhibitor Therapy for Cancer With Early Myocardial Tissue and Biomarker Changes During Treatment - Implication for Risk of Myocarditis and Cardiomyopathy
Brief Title: Immune Checkpoint Inhibitor Therapy for Cancer and Risk of Myocarditis or Cardiomyopathy
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Christian Houbois, Assistant Professor, MD, Sunnybrook Health Sciences Centre
Other Study IDs: 5993
Record Dates: First submitted 2024-02-12; First posted 2024-03-13 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Cardio-Oncology; Cardiomyopathy Due to Drug
Keywords: Cardio-Oncology; Immunotherapy; Cardiomyopathy; Cardiac MRI; Myocardial tissue changes
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with skin cancer eligible for dual ICI treatment.

SUMMARY:
Patients undergoing dual treatment with Immune checkpoint inhibitors (ICI) for various cancers, e.g. melanoma, are at increased risk of developing myocarditis and cardiomyopathy. Currently, only limited data on serial myocardial tissue changes during treatment and whether they predict outcomes are available. Cardiac MRI (CMR) is the reference standard for non-invasive myocardial volumes/function analysis and uniquely characterizes myocardial tissue. Therefore, it may help detect myocardial tissue changes during treatment and help early treatment and prevent adverse cardiac outcomes.

DETAILED DESCRIPTION:
As patients going through cancer therapy live longer, they are at a higher risk of developing cardiovascular disease. Hence the evolving field of Cardio-Oncology has garnered much attention and importance. In recent years, immune checkpoint inhibitors (ICI) have become an essential component of cancer therapy, significantly improving patient outcomes that were previously considered palliative, e.g. metastatic melanoma, renal cell or lung cancer, and these therapies have improved survival.

With ICI therapy and especially with combination therapy, patients may develop severe ICI-related adverse events, e.g. myocarditis (1-5%) which is fatal in 30-50% of the patients. Another more significant subgroup of patients will develop non-inflammatory cardiomyopathy or other major cardiac events like cardiovascular death, cardiac arrest etc. There is also evidence that during ICI treatment atherosclerotic disease may progress. Identifying patients at risk for both remains a major challenge and is a knowledge gap in Cardio-Oncology.

Cardiovascular magnetic resonance (CMR) is a unique, highly reproducible, multiparametric method for non-invasive myocardial tissue characterization for diagnosing myocardial inflammation. Biomarkers like quantitative cardiac relaxometry (T1/T2-Mapping) with extracellular volume fraction (ECV), delayed gadolinium enhancement (LGE) or myocardial strain show insights into myocardial tissue composition. These biomarkers have the potential to identify early myocardial changes before the risk of clinical myocarditis or non-inflammatory cardiomyopathy occurs and may therefore help identify early myocardial tissue changes during ICI treatment and help identify patients at risk early on. Also, CMR can assess the aorta with high temporal and spatial resolution to identify atherosclerotic changes.

Only a few retrospective studies and case reports with small numbers of patients have investigated ICI-related cardiac events during treatment. Evidence shows that many patients present with heart failure (~80%), but troponin is only elevated in ~45%. This indicates that ICI-associated left ventricular (LV) dysfunction may exist without troponin elevation. Other data suggests that the ICI-associated myocardial tissue inflammation pattern might differ from viral myocarditis. The myocardial T1/T2 relaxation times may be elevated during ICI-associated myocardial inflammation. There is also evidence that strain changes are associated with adverse events within 30 days of treatment. However, all these studies demonstrate CMR findings when patients have already developed LV dysfunction or myocarditis. The proposed project would be the first prospective study to get deeper insights into serial, systematic ICI-associated myocardial tissue changes during treatment and their correlation with serum biomarkers and clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age, or older, with skin cancer and eligible for ICI treatment with a combination of a) nivolumab, b) pembrolizumab, or c) ipilimumab.
* Able to provide informed consent
* Able to travel to SHSC for cardiac imaging.

Exclusion Criteria:

* Life expectancy equal to, or less than, 12 months
* Participating in another clinical trial
* Treated with ICI in the past
* History of cardiac disease (e.g. heart failure, myocardial infarction, atrial fibrillation, unstable angina)
* Pregnant patients
* Impaired renal function (GFR equal to, or less than, 30mL/min)
* Contraindications for MRI (e.g. pacemaker).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This pilot study will include 15 patients recruited from Odette Cancer Centre at Sunnybrook Health Sciences Center who have skin cancer and are eligible for immunotherapy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Define changes in CMR tissue and blood biomarkers during ICI treatment. | Baseline, 6 weeks and 6 months
  The following parameters are investigated to assess for underlying myocardial remodelling and/or inflammation during treatment with ICI.
  Left ventricular volumes in ml Left ventricular ejection fraction in percentage T1 Mapping: T1 relaxation time in milliseconds T2 Mapping: T2 relaxation time in milliseconds ECV = (1-hematocrit) × (Δ(1/T1myocardium)/Δ(1/T1blood)) in percentage Strain (GCS, GLS, GRS) reported as a percentage, formula =(Max Length-Initial Length)/Initial Length LGE is qualitatively described as categorical variables e.g. epicardial, mid-myocardial, subendocardial or transmural.
  LGE is quantified as mass in gram and as percentage of the LV mass. High sensitivity troponin 1 nanogram/ mL B-type natriuretic peptide (BNP) nanogram/L High sensitivity CRP in mg/L
Investigate associations between CMR imaging biomarkers and CMR-defined left ventricular ejection fraction. | Baseline, 6 weeks and 6 months
  This analysis is to determine if the biomarkers are associated with LVEF changes over time.
  Left ventricular volumes in ml Left ventricular ejection fraction in percentage T1 Mapping: T1 relaxation time in milliseconds T2 Mapping: T2 relaxation time in milliseconds ECV = (1-hematocrit) × (Δ(1/T1myocardium)/Δ(1/T1blood)) in percentage Strain (GCS, GLS, GRS) reported as a percentage, formula =(Max Length-Initial Length)/Initial Length LGE is qualitatively described as categorical variables e.g. epicardial, mid-myocardial, subendocardial or transmural.
  LGE is quantified as mass in gram and as percentage of the LV mass.
Investigate associations between serum biomarkers and CMR-defined left ventricular ejection fraction. | Baseline, 6 weeks and 6 months
  This analysis is to determine if blood biomarkers are associated with LVEF changes over time.
  High sensitivity troponin 1 nanogram/ mL B-type natriuretic peptide (BNP) nanogram/L High sensitivity CRP in mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Christian Houbois, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data with other researchers.

REFERENCES:
- [Background] Thavendiranathan P, Abdel-Qadir H, Fischer HD, Camacho X, Amir E, Austin PC, Lee DS. Breast Cancer Therapy-Related Cardiac Dysfunction in Adult Women Treated in Routine Clinical Practice: A Population-Based Cohort Study. J Clin Oncol. 2016 Jul 1;34(19):2239-46. doi: 10.1200/JCO.2015.65.1505. Epub 2016 Apr 18. PMID 27091709
- [Background] Postow MA, Callahan MK, Wolchok JD. Immune Checkpoint Blockade in Cancer Therapy. J Clin Oncol. 2015 Jun 10;33(17):1974-82. doi: 10.1200/JCO.2014.59.4358. Epub 2015 Jan 20. PMID 25605845
- [Background] Postow MA, Chesney J, Pavlick AC, Robert C, Grossmann K, McDermott D, Linette GP, Meyer N, Giguere JK, Agarwala SS, Shaheen M, Ernstoff MS, Minor D, Salama AK, Taylor M, Ott PA, Rollin LM, Horak C, Gagnier P, Wolchok JD, Hodi FS. Nivolumab and ipilimumab versus ipilimumab in untreated melanoma. N Engl J Med. 2015 May 21;372(21):2006-17. doi: 10.1056/NEJMoa1414428. Epub 2015 Apr 20. PMID 25891304
- [Background] Wang DY, Salem JE, Cohen JV, Chandra S, Menzer C, Ye F, Zhao S, Das S, Beckermann KE, Ha L, Rathmell WK, Ancell KK, Balko JM, Bowman C, Davis EJ, Chism DD, Horn L, Long GV, Carlino MS, Lebrun-Vignes B, Eroglu Z, Hassel JC, Menzies AM, Sosman JA, Sullivan RJ, Moslehi JJ, Johnson DB. Fatal Toxic Effects Associated With Immune Checkpoint Inhibitors: A Systematic Review and Meta-analysis. JAMA Oncol. 2018 Dec 1;4(12):1721-1728. doi: 10.1001/jamaoncol.2018.3923. PMID 30242316
- [Background] Lyon AR, Yousaf N, Battisti NML, Moslehi J, Larkin J. Immune checkpoint inhibitors and cardiovascular toxicity. Lancet Oncol. 2018 Sep;19(9):e447-e458. doi: 10.1016/S1470-2045(18)30457-1. PMID 30191849
- [Background] Escudier M, Cautela J, Malissen N, Ancedy Y, Orabona M, Pinto J, Monestier S, Grob JJ, Scemama U, Jacquier A, Lalevee N, Barraud J, Peyrol M, Laine M, Bonello L, Paganelli F, Cohen A, Barlesi F, Ederhy S, Thuny F. Clinical Features, Management, and Outcomes of Immune Checkpoint Inhibitor-Related Cardiotoxicity. Circulation. 2017 Nov 21;136(21):2085-2087. doi: 10.1161/CIRCULATIONAHA.117.030571. No abstract available. PMID 29158217
- [Background] Zhang L, Awadalla M, Mahmood SS, Nohria A, Hassan MZO, Thuny F, Zlotoff DA, Murphy SP, Stone JR, Golden DLA, Alvi RM, Rokicki A, Jones-O'Connor M, Cohen JV, Heinzerling LM, Mulligan C, Armanious M, Barac A, Forrestal BJ, Sullivan RJ, Kwong RY, Yang EH, Damrongwatanasuk R, Chen CL, Gupta D, Kirchberger MC, Moslehi JJ, Coelho-Filho OR, Ganatra S, Rizvi MA, Sahni G, Tocchetti CG, Mercurio V, Mahmoudi M, Lawrence DP, Reynolds KL, Weinsaft JW, Baksi AJ, Ederhy S, Groarke JD, Lyon AR, Fradley MG, Thavendiranathan P, Neilan TG. Cardiovascular magnetic resonance in immune checkpoint inhibitor-associated myocarditis. Eur Heart J. 2020 May 7;41(18):1733-1743. doi: 10.1093/eurheartj/ehaa051. PMID 32112560
- [Background] Drobni ZD, Gongora C, Taron J, Suero-Abreu GA, Karady J, Gilman HK, Supraja S, Nikolaidou S, Leeper N, Merkely B, Maurovich-Horvat P, Foldyna B, Neilan TG. Impact of immune checkpoint inhibitors on atherosclerosis progression in patients with lung cancer. J Immunother Cancer. 2023 Jul;11(7):e007307. doi: 10.1136/jitc-2023-007307. PMID 37433718
- [Background] Bellenger NG, Burgess MI, Ray SG, Lahiri A, Coats AJ, Cleland JG, Pennell DJ. Comparison of left ventricular ejection fraction and volumes in heart failure by echocardiography, radionuclide ventriculography and cardiovascular magnetic resonance; are they interchangeable? Eur Heart J. 2000 Aug;21(16):1387-96. doi: 10.1053/euhj.2000.2011. PMID 10952828
- [Background] Grothues F, Smith GC, Moon JC, Bellenger NG, Collins P, Klein HU, Pennell DJ. Comparison of interstudy reproducibility of cardiovascular magnetic resonance with two-dimensional echocardiography in normal subjects and in patients with heart failure or left ventricular hypertrophy. Am J Cardiol. 2002 Jul 1;90(1):29-34. doi: 10.1016/s0002-9149(02)02381-0. PMID 12088775
- [Background] Quinaglia T, Gongora C, Awadalla M, Hassan MZO, Zafar A, Drobni ZD, Mahmood SS, Zhang L, Coelho-Filho OR, Suero-Abreu GA, Rizvi MA, Sahni G, Mandawat A, Zatarain-Nicolas E, Mahmoudi M, Sullivan R, Ganatra S, Heinzerling LM, Thuny F, Ederhy S, Gilman HK, Sama S, Nikolaidou S, Mansilla AG, Calles A, Cabral M, Fernandez-Aviles F, Gavira JJ, Gonzalez NS, Garcia de Yebenes Castro M, Barac A, Afilalo J, Zlotoff DA, Zubiri L, Reynolds KL, Devereux R, Hung J, Picard MH, Yang EH, Gupta D, Michel C, Lyon AR, Chen CL, Nohria A, Fradley MG, Thavendiranathan P, Neilan TG. Global Circumferential and Radial Strain Among Patients With Immune Checkpoint Inhibitor Myocarditis. JACC Cardiovasc Imaging. 2022 Nov;15(11):1883-1896. doi: 10.1016/j.jcmg.2022.06.014. Epub 2022 Sep 14. PMID 36357131
- [Background] Mordi I, Carrick D, Bezerra H, Tzemos N. T1 and T2 mapping for early diagnosis of dilated non-ischaemic cardiomyopathy in middle-aged patients and differentiation from normal physiological adaptation. Eur Heart J Cardiovasc Imaging. 2016 Jul;17(7):797-803. doi: 10.1093/ehjci/jev216. Epub 2015 Sep 10. PMID 26358692
- [Background] Thavendiranathan P, Walls M, Giri S, Verhaert D, Rajagopalan S, Moore S, Simonetti OP, Raman SV. Improved detection of myocardial involvement in acute inflammatory cardiomyopathies using T2 mapping. Circ Cardiovasc Imaging. 2012 Jan;5(1):102-10. doi: 10.1161/CIRCIMAGING.111.967836. Epub 2011 Oct 28. PMID 22038988
- [Background] Messroghli DR, Moon JC, Ferreira VM, Grosse-Wortmann L, He T, Kellman P, Mascherbauer J, Nezafat R, Salerno M, Schelbert EB, Taylor AJ, Thompson R, Ugander M, van Heeswijk RB, Friedrich MG. Clinical recommendations for cardiovascular magnetic resonance mapping of T1, T2, T2* and extracellular volume: A consensus statement by the Society for Cardiovascular Magnetic Resonance (SCMR) endorsed by the European Association for Cardiovascular Imaging (EACVI). J Cardiovasc Magn Reson. 2017 Oct 9;19(1):75. doi: 10.1186/s12968-017-0389-8. PMID 28992817
- [Background] Hor KN, Gottliebson WM, Carson C, Wash E, Cnota J, Fleck R, Wansapura J, Klimeczek P, Al-Khalidi HR, Chung ES, Benson DW, Mazur W. Comparison of magnetic resonance feature tracking for strain calculation with harmonic phase imaging analysis. JACC Cardiovasc Imaging. 2010 Feb;3(2):144-51. doi: 10.1016/j.jcmg.2009.11.006. PMID 20159640
- [Background] Sawaya H, Sebag IA, Plana JC, Januzzi JL, Ky B, Cohen V, Gosavi S, Carver JR, Wiegers SE, Martin RP, Picard MH, Gerszten RE, Halpern EF, Passeri J, Kuter I, Scherrer-Crosbie M. Early detection and prediction of cardiotoxicity in chemotherapy-treated patients. Am J Cardiol. 2011 May 1;107(9):1375-80. doi: 10.1016/j.amjcard.2011.01.006. Epub 2011 Mar 2. PMID 21371685
- [Background] Nakano S, Takahashi M, Kimura F, Senoo T, Saeki T, Ueda S, Tanno J, Senbonmatsu T, Kasai T, Nishimura S. Cardiac magnetic resonance imaging-based myocardial strain study for evaluation of cardiotoxicity in breast cancer patients treated with trastuzumab: A pilot study to evaluate the feasibility of the method. Cardiol J. 2016;23(3):270-80. doi: 10.5603/CJ.a2016.0023. Epub 2016 May 13. PMID 27173679
- [Background] Cadour F, Cautela J, Rapacchi S, Varoquaux A, Habert P, Arnaud F, Jacquier A, Meilhac A, Paganelli F, Lalevee N, Scemama U, Thuny F. Cardiac MRI Features and Prognostic Value in Immune Checkpoint Inhibitor-induced Myocarditis. Radiology. 2022 Jun;303(3):512-521. doi: 10.1148/radiol.211765. Epub 2022 Mar 1. PMID 35230185
- [Background] Thavendiranathan P, Zhang L, Zafar A, Drobni ZD, Mahmood SS, Cabral M, Awadalla M, Nohria A, Zlotoff DA, Thuny F, Heinzerling LM, Barac A, Sullivan RJ, Chen CL, Gupta D, Kirchberger MC, Hartmann SE, Weinsaft JW, Gilman HK, Rizvi MA, Kovacina B, Michel C, Sahni G, Gonzalez-Mansilla A, Calles A, Fernandez-Aviles F, Mahmoudi M, Reynolds KL, Ganatra S, Gavira JJ, Gonzalez NS, Garcia de Yebenes Castro M, Kwong RY, Jerosch-Herold M, Coelho-Filho OR, Afilalo J, Zatarain-Nicolas E, Baksi AJ, Wintersperger BJ, Calvillo-Arguelles O, Ederhy S, Yang EH, Lyon AR, Fradley MG, Neilan TG. Myocardial T1 and T2 Mapping by Magnetic Resonance in Patients With Immune Checkpoint Inhibitor-Associated Myocarditis. J Am Coll Cardiol. 2021 Mar 30;77(12):1503-1516. doi: 10.1016/j.jacc.2021.01.050. PMID 33766256
- [Background] Schulz-Menger J, Bluemke DA, Bremerich J, Flamm SD, Fogel MA, Friedrich MG, Kim RJ, von Knobelsdorff-Brenkenhoff F, Kramer CM, Pennell DJ, Plein S, Nagel E. Standardized image interpretation and post-processing in cardiovascular magnetic resonance - 2020 update : Society for Cardiovascular Magnetic Resonance (SCMR): Board of Trustees Task Force on Standardized Post-Processing. J Cardiovasc Magn Reson. 2020 Mar 12;22(1):19. doi: 10.1186/s12968-020-00610-6. PMID 32160925